CLINICAL TRIAL: NCT02595918
Title: A Pilot Study of Preoperative Nivolumab in High-Risk Non-Metastatic and Metastatic Renal Cell Carcinoma
Brief Title: Nivolumab in Treating Patients With High-Risk Kidney Cancer Before Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01913; NCI-2015-01913 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-195; 16-195 A(1); 9913 (Other: Memorial Sloan Kettering Cancer Center); 9913 (Other: CTEP); P30CA008748 (NIH)
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Clear Cell Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Stage I Renal Cell Cancer AJCC v6 and v7; Stage II Renal Cell Cancer AJCC v7; Stage III Renal Cell Cancer AJCC v7; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Metastasectomy; Nephrectomy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes on days -56, -42, -28, and -14 in the absence of disease progression or unacceptable toxicity. Patients then undergo nephrectomy or metastasectomy on day 0.
  Interventions: Procedure: Metastasectomy; Procedure: Nephrectomy; Biological: Nivolumab

INTERVENTIONS:
Procedure: Metastasectomy — Undergo metastasectomy
Procedure: Nephrectomy — Undergo nephrectomy
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This pilot phase I trial studies the side effects of nivolumab and how well it works in treating patients with high-risk kidney cancer before surgery. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To study the safety and feasibility of preoperative nivolumab administration in subjects with resectable, high-risk, non-metastatic and metastatic renal cell carcinoma undergoing planned cytoreductive nephrectomy or metastasectomy.

SECONDARY OBJECTIVES:

I. To assess overall response rate in patients receiving preoperative nivolumab.

II. To assess recurrence free survival at 2 years in patients receiving preoperative nivolumab in patients with high-risk, non-metastatic disease.

EXPLORATORY OBJECTIVES:

I. To evaluate the association between baseline tumor mutational burden and both immune infiltration and radiographic tumor response to nivolumab.

II. To explore predicted and expressed tumor neoantigens and their correlation with radiographic tumor response to nivolumab.

III. To explore the association between the predicted immune signature (via ribonucleic acid sequencing [RNAseq]) in the tumor microenvironment with radiographic tumor response to nivolumab.

IV. To determine whether changes in the tumor microenvironment before, during, and after therapy are associated with response.

V. To assess the potential association between PD-L1 expression (by immunohistochemistry [IHC]) and radiographic tumor response to nivolumab.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on days -56, -42, -28, and -14 in the absence of disease progression or unacceptable toxicity. Patients then undergo nephrectomy or metastasectomy on day 0.

After completion of study treatment, patients are followed up at 14-28 days, at 90 days, and then at 24-28 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed clear cell renal cell carcinoma (RCC)
* For non-metastatic patients, the preoperative Memorial Sloan-Kettering (MSK) nomogram estimates the patient's likelihood of freedom from metastatic recurrence within the first 12 years following radical or partial nephrectomy to be =< 80%
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Non-metastatic disease will be defined by no evidence of metastases other than regional lymphadenopathy as assessed by imaging of the chest, abdomen and pelvis with CT of the chest and CT or MRI of the abdomen; regional lymph nodes, per 7th edition American Joint Committee on Cancer (AJCC) staging manual (2010) for kidney cancer, include the following positions: renal hilar, precaval, paracaval, retrocaval, interaortocaval, paraaortic, preaortic, and retroaortic
* Scheduled to undergo nephrectomy or metastasectomy as part of treatment plan, per assessment through an MSK urologic surgeon or medical oncologist listed as investigator on this trial
* Availability of a frozen biopsy core prior to cycle 1, day 1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Karnofsky >= 80%)
* Leukocytes >= 2,500/mcL
* Absolute neutrophil count >= 1,500/mcL (without granulocyte colony-stimulating factor support within 2 weeks prior to cycle 1, day 1)
* Platelets >= 100,000/mcL (without transfusion within 2 weeks prior to cycle 1, day 1)
* Hemoglobin >= 9.0 g/dL (patients may be transfused to meet this criterion)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (except patients with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Creatinine =< 1.5 x ULN OR creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula)
* The effects of nivolumab on the developing human fetus are unknown; for this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; WOCBP should use an adequate method to avoid pregnancy for 23 weeks after the last dose of investigational drug; women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 14 days prior to the start of nivolumab; women must not be breastfeeding; men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception
* Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level greater than 40 mIU/mL
* WOCBP receiving nivolumab will be instructed to adhere to contraception for a period of 23 weeks after the last dose of investigational product; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; these durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days and men who are sexually active with WOCBP use contraception for 5 half-lives plus 90 days
* Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior receipt of systemic checkpoint inhibitor therapy for renal cell carcinoma
* Inability to safely delay surgery by 8 weeks as per surgeon's discretion
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab
* History of severe hypersensitivity reaction to any monoclonal antibody
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because nivolumab has a potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab, breastfeeding should be discontinued if the mother is treated with nivolumab
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Patients should be excluded if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome, psoriasis controlled with topical medication, and patients with positive serology, such as antinuclear antibodies (ANA) or anti-thyroid antibodies, should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of study drug administration; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Diagnosis of any second malignancy within the last 5 years prior to cycle 1, day 1, with the exception of those with a negligible risk of metastasis or death, per investigator's discretion (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
* Use of live vaccines against infectious disease (e.g. varicella) within 28 days of initiation of study therapy; killed vaccinations (e.g. influenza) are allowed at any appropriate time before and during the study
* Life expectancy < 3 months, per consenting investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of a patient to receive at least 3 doses of nivolumab and complete surgery without significant delay attributable to nivolumab therapy | Up to 8 weeks
  Significant delay is defined as delay of > 112 days after the first dose of nivolumab, which would constitute a doubling of the 'planned delay' that our design requires for administration of preoperative therapy (56 days).

SECONDARY OUTCOMES:
Incidence of toxicity | Up to 90 days
  Will be defined per Common Terminology Criteria for Adverse Events version 4.0 (version 5.0 beginning April 1, 2018). All patients who receive any amount of the study drug will be evaluable for toxicity. Toxicity will be summarized according to grade as a number and percentage of participants. Each adverse event will be summarized as the highest grade experienced for an individual patient. Descriptive statistics will be used for summaries of the reported toxicity.
Surgical complications | Up to 90 days
  Defined per Clavien-Dindo Complications score.
Overall response rate | Up to 2 years
  Will be measured by radiographic response assessment for each cross sectional scan obtained using Response Evaluation Criteria in Solid Tumors 1.1. All patients will be categorized per their best radiographic response (complete response/partial response/stable disease/progressive disease), and the frequency of each category will be determined. The overall response rate will be calculated by dividing the sum of all patients achieving a complete response or confirmed partial response by the number of all evaluable patients.
Recurrence free survival | Time from the start of the treatment to recurrence or death, assessed up to 2 years
  Recurrence free survival will be estimated using the Kaplan-Meier method. Two-year recurrence free survival will be provided along with 95% confidence interval. Patients who are unable to undergo nephrectomy or metastasectomy for any reason will not be included in the analysis.

OTHER OUTCOMES:
Feasibility of biomarker analysis | Up to 90 days
  Will be defined as ability to procure sufficient quantity and quality of tumor tissue and peripheral blood for testing. Will be descriptive or graphical in nature, and are designed to generate new hypotheses to be tested in future clinical studies. When parameters of immune response are measured, continuous variables will be summarized with means and standard deviations. Dichotomous and categorical variables will be summarized using proportions with exact 95% confidence intervals and counts, respectively. For each patient, comparisons in the pre and post-nivolumab responses will be compared using paired t-tests (or Wilcoxon signed rank tests if appropriate) for continuous variables.

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Voss, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Golkaram M, Kuo F, Gupta S, Carlo MI, Salmans ML, Vijayaraghavan R, Tang C, Makarov V, Rappold P, Blum KA, Zhao C, Mehio R, Zhang S, Godsey J, Pawlowski T, DiNatale RG, Morris LGT, Durack J, Russo P, Kotecha RR, Coleman J, Chen YB, Reuter VE, Motzer RJ, Voss MH, Liu L, Reznik E, Chan TA, Hakimi AA. Spatiotemporal evolution of the clear cell renal cell carcinoma microenvironment links intra-tumoral heterogeneity to immune escape. Genome Med. 2022 Dec 19;14(1):143. doi: 10.1186/s13073-022-01146-3. PMID 36536472